CLINICAL TRIAL: NCT01442441
Title: How Pathologic Features of Chronic Pancreatitis Corelate With Endoscopic Ultrasound (EUS) Criteria for Diagnosing Chronic Pancreatitis
Brief Title: Correlation of Chronic Pancreatitis Pathology Features With Endoscopic Ultrasound (EUS) Criteria
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Other Study IDs: 0809-67
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Pancreatitis
Keywords: chronic pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic pancreatitis

SUMMARY:
In this research project the investigators intend to find out if Endoscopic Ultrasound (EUS) criteria for diagnosing chronic pancreatitis can be correlated with pathologic characteristics of tissues taken from pancreas of patients with suspected chronic pancreatitis.

This will be a retrospective study which will examine results from biopsy specimens and endoscopic ultrasound findings in suspected chronic pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* will include all patients who consented to have both EUS and had biopsy taken for tissue diagnosis.

Exclusion Criteria:

* Will exclude patients who are less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Retrospective surgery cases who had chronic pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-02; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States